CLINICAL TRIAL: NCT02671084
Title: Effect of Sevoflurane on CKMB Release After PCI With Drug-eluting Stents: a Randomised Trial
Brief Title: Sevoflurane and Percutaneous Coronary Intervention by Stent
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: interim analysis suggests futility
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, RONALDO ROSSI JUNIOR, Principal Investigator, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 090106/2015
Record Dates: First submitted 2016-01-20; First posted 2016-02-02 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Myocardial Infarction
Keywords: Sevoflurane; Ck-MB
MeSH Terms: conditions — Myocardial Infarction | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Sevoflurane Group (Experimental): Sevoflurane Group called group A patients will receive sevoflurane. The patients of group A will receive facial mask properly attached to your face, inspiratory fraction of sevoflurane 3%, with therapeutic target of 1.2% expired fraction into spontaneously breathing.This exposure will during 30 min. Than, the mask will remove of the face and the patient will spontaneously breathing in ambient air during 10 min. This procedure is sufficient to induce the pre anesthetic conditioning in the group exposed to sevoflurane. After the end of this exhibition, patients will be allowed to enter the catheterization laboratory for angioplasty, no more any anesthetic agent will be administer until the end of his procedure.
  Interventions: Drug: sevoflurane
- Control Group (Placebo Comparator): Control Group called group B patients who will not receive sevoflurane. The patient of group B will receive facial mask properly attached to your face into spontaneously breathing.This exposure will during 30 min. Than, the mask will remove of the face and the patient will spontaneously breathing in ambient air during 10 min. After the end of this exhibition, patients will be allowed to enter the catheterization laboratory for angioplasty, no more any anesthetic agent will be administer until the end of his procedure.
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: sevoflurane — compare effect of sevoflurane when administered before PCI

SUMMARY:
Increase in CK-MB after percutaneous coronary angioplasty more than 100% of baseline can represents a problem to the patients resulting in increase of morbidity and mortality.

Patients submitted of coronary angioplasty procedures can release in varying degrees of creatine kinase, MB isoform (CK - MB), on the order of 30% of all angioplasty.

Possibly patients who will receive sevoflurane experience a higher level of cardiac cell protection with lower incidence in the release of CK - MB values in excess of 100% baseline.

DETAILED DESCRIPTION:
Several published clinical studies have shown the benefit of using inhaled anesthetic agents in patients undergoing coronary artery bypass graft(CABG). These benefits involve functional state of the heart and reduction damage to the organ. These events are related to intracellular phenomena that result in intracellular calcium homeostasis giving physical and functional benefits to the heart. Also disclosed is a modulation of the inflammatory response to endothelial level with resulting protective character to the coronary bed.

Patients submitted of coronary angioplasty procedures can release in varying degrees of creatine kinase, MB isoform (CK - MB), on the order of 30% of all angioplasty. Even in smaller increases than 3 times baseline, a criterion that defines myocardial infarction, clinical impact can already be found. Increase in CK-MB more than 100% of baseline can represents a problem to the patients. This elevation of CK - MB is associated with various factors such as age, characteristic of the lesion, clinical status of the patient, inferring that endovascular procedures of coronary, simple or complex, have associated myocardial damage, which depending on the intensity of the damage, results in increased morbidity and mortality.

BACKGROUND AND OBJECTIVES:

Check for reduction in the percentage of patients that release CK -MB at levels above the 100% baseline in patients anesthetized with sevoflurane compared to the control group. Possibly patients who will receive sevoflurane experience a higher level of cardiac cell protection with lower incidence in the release of CK - MB values in excess of 100% baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Both gender.
2. Patients with coronary artery disease candidates for coronary angioplasty stent.
3. Cardiac catheterization on an urgent basis.
4. Coronary angioplasty in elective and urgency.
5. Age less than 80 years.

Exclusion Criteria:

1. Patients aged greater than or equal of 80 years.
2. Angioplasty balloon catheter statement.
3. Myocardial infarction with ST-segment elevation.
4. Angioplasty in saphenous vein grafts in patients after surgical revascularization.
5. Patient pregnant.
6. Dialytic insufficiency renal.
7. Patients submited a urgent cardiac catheterization but not progress with coronary angioplasty stent.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Measure level of Ck-MB in all patients | 24 hours after coronary intervention

SECONDARY OUTCOMES:
Length of stay in hospital | 30 days after coronary intervention
  It will be quantified the length of hospital stay of patients who underwent coronary intervention checking if there is difference between groups
Length of stay in Intensive Care Unit (UCI) | 30 days after coronary intervention
  The length of stay in UCI will be quantified if patients who underwent coronary intervention are referred to this sector
mortality rate | 1 year after coronary intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Dante Pazzanese of Cardiology, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in journals
Supporting Information: Study Protocol

REFERENCES:
- [Result] Landoni G, Zangrillo A, Fochi O, Maj G, Scandroglio AM, Morelli A, Tritapepe L, Montorfano M, Colombo A. Cardiac protection with volatile anesthetics in stenting procedures. J Cardiothorac Vasc Anesth. 2008 Aug;22(4):543-7. doi: 10.1053/j.jvca.2008.02.020. Epub 2008 May 14. PMID 18662628
- [Result] Jang JS, Jin HY, Seo JS, Yang TH, Kim DK, Kim DS, Cho KI, Kim BH, Je HG, Park YH. Prognostic value of creatine kinase-myocardial band isoenzyme elevation following percutaneous coronary intervention: a meta-analysis. Catheter Cardiovasc Interv. 2013 May;81(6):959-67. doi: 10.1002/ccd.24542. Epub 2012 Nov 14. PMID 22744792
- [Result] Lavi S, Alemayehu M, McCarty D, Warrington J, Lavi R. One-year outcome of the sevoflurane in acute myocardial infarction randomized trial. Can J Anaesth. 2015 Dec;62(12):1279-86. doi: 10.1007/s12630-015-0456-2. Epub 2015 Aug 22. PMID 26296299
- See also: Cardiac protection with volatile anesthetics in stenting procedures. — https://www.ncbi.nlm.nih.gov/pubmed/18662628
- See also: Prognostic value of creatine kinase-myocardial band isoenzyme elevation following percutaneous coronary intervention: a meta-analysis. — http://www.ncbi.nlm.nih.gov/pubmed/22744792
- See also: One-year outcome of the sevoflurane in acute myocardial infarction randomized trial. — http://www.ncbi.nlm.nih.gov/pubmed/26296299